CLINICAL TRIAL: NCT05245929
Title: Evaluation of Two Bone Anchored Appliances for en Masse Distalization of Maxillary Buccal Segment in Class II Patients: A Comparative Clinical Study
Brief Title: En Masse Distaliaztion Via Skeletal Anchorage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Kadry Ahmed Algariah, Research Assistant, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dist007
Record Dates: First submitted 2022-02-09; First posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Orthodontic Appliance Complication, Angle Class II Patients, Distalization

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Skeletally anchored Distal Jet appliance (Active Comparator)
  Interventions: Device: Distalization
- Skeletally anchored Hyrax screw distalizer (Active Comparator)
  Interventions: Device: Distalization

INTERVENTIONS:
Device: Distalization — Distalizing the posterior maxillary segment

SUMMARY:
Comparing the efficacy and performance of two conventionally anchored distalizers after modifying them to be skeletally anchored. En masse distalization is attempted by consolidating the posterior maxillary segment "first premolar to second molar" as one unit.

ELIGIBILITY:
Inclusion Criteria:

* Full set of permanent teeth present, except for third molar
* Bilateral Class II malocclusion with a mesial migration of maxillary posterior teeth
* No systemic conditions interfering with treatment, as reported by patient
* No previous Orthodontic treatment
* Good Oral Hygiene
* No use of any for of anti-inflammatory drugs

Exclusion Criteria:

* Patient who required surgery to correct skeletal discrepancies
* Patient with congenital dentoskeletal disorders
* Missed or Mutilated teeth in Maxillary arch
* Patients with poor oral hygiene

Ages: 14 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2021-01-05 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Amount of distalization | 6 months
  difference in initial and final position of maxillary posterior segment

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar University, faculty of dental medicine orthodontic clinic, Cairo, Nasr City, Egypt

IPD SHARING:
Plan to Share IPD: Undecided